CLINICAL TRIAL: NCT06161571
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety and Efficacy of Efruxifermin in Subjects With Non-invasively Diagnosed Nonalcoholic Steatohepatitis (NASH)/Metabolic Dysfunction-Associated Steatohepatitis (MASH) and Nonalcoholic Fatty Liver Disease (NAFLD)/Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD)
Brief Title: A Study Evaluating Efruxifermin in Subjects With Non-invasively Diagnosed Nonalcoholic Steatohepatitis (NASH)/Metabolic Dysfunction-Associated Steatohepatitis (MASH) and Nonalcoholic Fatty Liver Disease (NAFLD)/Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Akero Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK-US-001-0107
Record Dates: First submitted 2023-11-22; First posted 2023-12-08 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-06

CONDITIONS: NASH/MASH; NAFLD/MASLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- EFX 50 mg (Experimental)
  Interventions: Drug: Efruxifermin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- EFX 50 mg (Open-Label Rollover) (Experimental)
  Interventions: Drug: Efruxifermin

INTERVENTIONS:
Drug: Efruxifermin — Administered by subcutaneous (SC) injection
  Arms: EFX 50 mg; EFX 50 mg (Open-Label Rollover)
Drug: Placebo — Administered by SC injection
  Arms: Placebo

SUMMARY:
The aim of this study is to assess the safety and tolerability of EFX compared to placebo in subjects with non-invasively diagnosed NASH/MASH and NAFLD/MASLD.

ELIGIBILITY:
Inclusion Criteria:

Main Study Only:

* Males and non-pregnant, non-lactating females between 18 - 80 (between 19-80 in the Republic of Korea) years of age inclusive, on the day of signing informed consent
* Previous history or presence of 2 out of 4 components of metabolic syndrome (obesity, dyslipidemia, elevated blood pressure, elevated fasting glucose) or type 2 diabetes
* Suspected or confirmed diagnosis of NASH/MASH or NAFLD/MASLD or non-invasively diagnosed NASH/MASH or NAFLD/MASLD

Open-Label Rollover

* Prior participation in a previous Akero Phase 2 study

Exclusion Criteria:

* Other causes of liver disease based on medical history and/or liver histology and/or central laboratory results, including but not limited to: alcoholic liver disease, autoimmune disorders (e.g., primary biliary cholangitis [PBC], primary sclerosing cholangitis [PSC], autoimmune hepatitis), drug induced hepatotoxicity, Wilson disease, clinically significant iron overload, or alpha-1-antitrypsin deficiency
* Type 1 or unstable Type 2 diabetes

A reduced list of inclusion and exclusion criteria apply to participants in the open-label rollover extension.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Extent of exposure | 52 Weeks
  A participant's extent of exposure to study drug (weeks) will be generated from the data recorded in the study drug administration eCRF.
Number of participants with adverse events | 52 Weeks
  An adverse event (AE) is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug, whether or not related to the study drug.
Number of participants with adverse events by severity | 52 Weeks
  All AEs, both serious and non-serious, will be assessed for severity using the Common Terminology Criteria for Adverse Events v5.0.
Number of participants with clinically significant changes in clinical assessments | 52 Weeks
  Clinical assessments include clinical laboratory tests, electrocardiogram, ultrasounds, vital sign assessments, and concomitant medication usage.

SECONDARY OUTCOMES:
Percentage of participants with reduction in enhanced liver fibrosis (ELF) score by ≥ 0.5 and reduction in liver stiffness measurement (LSM) by ≥ 30% | 52 Weeks
Change from baseline in non-invasive marker ELF score | 52 Weeks
  ELF scale of 6.7 to 9.8 where higher scores indicative of increased fibrosis.
Change from baseline in non-invasive marker pro-peptide of type 3 procollagen (Pro-C3) | 52 Weeks
Change from baseline in non-invasive marker liver stiffness assessed by transient elastography (kPa, CAP) | 52 Weeks
Percentage of participants with a reduction in ELF score by ≥ 0.5 | 52 Weeks
Percentage of participants with a reduction in LSM by ≥ 30% | 52 Weeks
Change from baseline in lipoproteins | 52 Weeks
  Total cholesterol (mg/dL), Triglycerides (TG) (mg/dL), high density lipoprotein cholesterol (HDL-C) (mg/dL), Non-HDL-C (mg/dL), and low-density lipoprotein cholesterol (LDL-C) (mg/dL).
Change from baseline in markers of glycemic control: HbA1c (%) | 52 Weeks
Change from baseline in markers of glycemic control: adiponectin (mg/L) | 52 Weeks
Change from baseline in markers of liver injury | 52 Weeks
  Alanine aminotransferase (ALT) (U/L), aspartate aminotransferase (AST) (U/L), and gamma glutamyl transferase (GGT) (U/L).
Change from baseline in markers of liver injury: uric acid (mg/dL) | 52 Weeks
Change from baseline in body weight (kg) | 52 Weeks

CONTACTS AND LOCATIONS:
Locations (183):
- United States (120):
  - Akero Clinical Study Site, Birmingham, Alabama
  - Akero Clinical Study Site, Chandler, Arizona
  - Akero Clinical Study Site, Flagstaff, Arizona
  - Akero Clinical Study Site, Peoria, Arizona
  - Akero Clinical Study Site, Tucson, Arizona
  - Akero Clinical Study Site, Conway, Arkansas
  - Akero Clinical Study Site, Jonesboro, Arkansas
  - Akero Clinical Study Site, Little Rock, Arkansas
  - Akero Clinical Study Site, North Little Rock, Arkansas
  - Akero Clinical Study Site, Chula Vista, California
  - Akero Clinical Study Site, Coronado, California
  - Akero Clinical Study Site, Cypress, California
  - Akero Clinical Study Site, Inglewood, California
  - Akero Clinical Study Site, La Mesa, California
  - Akero Clinical Study Site, Lancaster, California
  - Akero Clinical Study Site, Los Angeles, California
  - Akero Clinical Study Site, Palm Springs, California
  - Akero Clinical Study Site, San Diego, California
  - Akero Clinical Study Site, San Francisco, California
  - Akero Clinical Study Site, Santa Maria, California
  - Akero Clinical Study Site, Englewood, Colorado
  - Akero Clinical Study Site, Bradenton, Florida
  - Akero Clinical Study Site, Brandon, Florida
  - Akero Clinical Study Site, Fort Myers, Florida
  - Akero Clinical Study Site, Gainesville, Florida
  - Akero Clinical Study Site, Hialeah Gardens, Florida
  - Akero Clinical Study Site, Inverness, Florida
  - Akero Clinical Study Site, Jacksonville, Florida
  - Akero Clinical Study Site, Lady Lake, Florida
  - Akero Clinical Study Site, Lakewood Rch, Florida
  - Akero Clinical Study Site, Largo, Florida
  - Akero Clinical Study Site, Maitland, Florida
  - Akero Clinical Study Site, Miami, Florida
  - Akero Clinical Study Site, Miami Lakes, Florida
  - Akero Clinical Study Site, Naples, Florida
  - Akero Clinical Study Site, Ocala, Florida
  - Akero Clinical Study Site, Port Orange, Florida
  - Akero Clinical Study Site, Sarasota, Florida
  - Akero Clinical Study Site, The Villages, Florida
  - Akero Clinical Study Site, Venice, Florida
  - Akero Clinical Study Site, Viera, Florida
  - Akero Clinical Study Site, West Palm Beach, Florida
  - Akero Clinical Study Site, Winter Park, Florida
  - Akero Clinical Study Site, Columbus, Georgia
  - Akero Clinical Study Site, Gainesville, Georgia
  - Akero Clinical Study Site, Marietta, Georgia
  - Akero Clinical Study Site, South Bend, Indiana
  - Akero Clinical Study Site, West Des Moines, Iowa
  - Akero Clinical Study Site, Topeka, Kansas
  - Akero Clinical Study Site, Wichita, Kansas
  - Akero Clinical Study Site, Bastrop, Louisiana
  - Akero Clinical Study Site, Covington, Louisiana
  - Akero Clinical Study Site, Houma, Louisiana
  - Akero Clinical Study Site, Marrero, Louisiana
  - Akero Clinical Study Site, Metairie, Louisiana
  - Akero Clinical Study Site, New Orleans, Louisiana
  - Akero Clinical Study Site, Shreveport, Louisiana
  - Akero Clinical Study Site, Baltimore, Maryland
  - Akero Clinical Study Site, Glen Burnie, Maryland
  - Akero Clinical Study Site, Greenbelt, Maryland
  - Akero Clinical Study Site, South Dartmouth, Massachusetts
  - Akero Clinical Study Site, Southfield, Michigan
  - Akero Clinical Study Site, Wyoming, Michigan
  - Akero Clinical Study Site, Ypsilanti, Michigan
  - Akero Clinical Study Site, Columbia, Missouri
  - Akero Clinical Study Site, Kansas City, Missouri
  - Akero Clinical Study Site, Las Vegas, Nevada
  - Akero Clinical Study Site, Reno, Nevada
  - Akero Clinical Study Site, Brick, New Jersey
  - Akero Clinical Study Site, Florham Park, New Jersey
  - Akero Clinical Study Site, Somers Point, New Jersey
  - Akero Clinical Study Site, Sparta, New Jersey
  - Akero Clinical Study Site, Santa Fe, New Mexico
  - Akero Clinical Study Site, New York, New York
  - Akero Clinical Study Site, Chapel Hill, North Carolina
  - Akero Clinical Study Site, Charlotte, North Carolina
  - Akero Clinical Study Site, Fayetteville, North Carolina
  - Akero Clinical Study Site, Morehead City, North Carolina
  - Akero Clinical Study Site, New Bern, North Carolina
  - Akero Clinical Study Site, Raleigh, North Carolina
  - Akero Clinical Study Site, Statesville, North Carolina
  - Akero Clinical Study Site, Columbus, Ohio
  - Akero Clinical Study Site, Dayton, Ohio
  - Akero Clinical Study Site, Springboro, Ohio
  - Akero Clinical Study Site, Westlake, Ohio
  - Akero Clinical Study Site, Philadelphia, Pennsylvania
  - Akero Clinical Study Site, Pittsburgh, Pennsylvania
  - Akero Clinical Study Site, Columbia, South Carolina
  - Akero Clinical Study Site, Summerville, South Carolina
  - Akero Clinical Study Site, Chattanooga, Tennessee
  - Akero Clinical Study Site, Clarksville, Tennessee
  - Akero Clinical Study Site, Hermitage, Tennessee
  - Akero Clinical Study Site, Nashville, Tennessee
  - Akero Clinical Study Site, Amarillo, Texas
  - Akero Clinical Study Site, Austin, Texas
  - Akero Clinical Study Site, Bellaire, Texas
  - Akero Clinical Study Site, Brownsville, Texas
  - Akero Clinical Study Site, Corpus Christi, Texas
  - Akero Clinical Study Site, Dallas, Texas
  - Akero Clinical Study Site, Edinburg, Texas
  - Akero Clinical Study Site, Fort Worth, Texas
  - Akero Clinical Study Site, Houston, Texas
  - Akero Clinical Study Site, Lewisville, Texas
  - Akero Clinical Study Site, McAllen, Texas
  - Akero Clinical Study Site, San Antonio, Texas
  - Akero Clinical Study Site, San Marcos, Texas
  - Akero Clinical Study Site, Waco, Texas
  - Akero Clinical Study Site, Webster, Texas
  - Akero Clinical Study Site, Wichita Falls, Texas
  - Akero Clinical Study Site, Ogden, Utah
  - Akero Clinical Study Site, Salt Lake City, Utah
  - Akero Clinical Study Site, Sandy City, Utah
  - Akero Clinical Study Site, South Ogden, Utah
  - Akero Clinical Study Site, Falls Church, Virginia
  - Akero Clinical Study Site, Norfolk, Virginia
  - Akero Clinical Study Site, Richmond, Virginia
  - Akero Clinical Study Site, Roanoke, Virginia
  - Akero Clinical Study Site, Suffolk, Virginia
  - Akero Clinical Study Site, Seattle, Washington
  - Akero Clinical Study Site, Spokane, Washington
- Argentina (3):
  - Akero Clinical Study Site, Ramos Mejía, Buenos Aires
  - Akero Clinical Study Site, Buenos Aires, Distrito Federal
  - Akero Clinical Study Site, Buenos Aires
- Australia (9):
  - Akero Clinical Study Site, Broadmeadow, New South Wales
  - Akero Clinical Study Site, Westmead, New South Wales
  - Akero Clinical Study Site, Adelaide, South Australia
  - Akero Clinical Study Site, Clayton, Victoria
  - Akero Clinical Study Site, Epping, Victoria
  - Akero Clinical Study Site, Heidelberg, Victoria
  - Akero Clinical Study Site, Melbourne, Victoria
  - Akero Clinical Study Site, Murdoch, Western Australia
  - Akero Clinical Study Site, Perth, Western Australia
- Canada (5):
  - Akero Clinical Study Site, Edmonton, Alberta
  - Akero Clinical Study Site, Hamilton, Ontario
  - Akero Clinical Study Site, Toronto, Ontario
  - Akero Clinical Study Site, Vaughan, Ontario
  - Akero Clinical Study Site, Terrebonne, Quebec
- India (14):
  - Akero Clinical Study Site, Surat, Gujarat
  - Akero Clinical Study Site, Vadodara, Gujarat
  - Akero Clinical Study Site, Thiruvananthapuram, Kerala
  - Akero Clinical Study Site, Dahegaon, Maharashtra
  - Akero Clinical Study Site, Mumbai, Maharashtra
  - Akero Clinical Study Site, Nagpur, Maharashtra
  - Akero Clinical Study Site, Pune, Maharashtra
  - Akero Clinical Study Site, New Delhi, National Capital Territory of Delhi
  - Akero Clinical Study Site, Chandigarh, Punjab
  - Akero Clinical Study Site, Jaipur, Rajasthan
  - Akero Clinical Study Site, Coimbatore, Tamil Nadu
  - Akero Clinical Study Site, Hyderabad, Telangana
  - Akero Clinical Study Site, Varanasi, Uttar Pradesh
  - Akero Clinical Study Site, Kolkata, West Bengal
- Israel (8):
  - Akero Clinical Study Site, Petah Tikva, Central District
  - Akero Clinical Study Site, Ramat Gan, Central District
  - Akero Clinical Study Site, Haifa, Haifa District
  - Akero Clinical Study Site, Afula, Northern District
  - Akero Clinical Study Site, Nahariya, Northern District
  - Akero Clinical Study Site, Nazareth, Northern District
  - Akero Clinical Study Site, Jerusalem
  - Akero Clinical Study Site, Tel Aviv
- Akero Clinical Study Site, Mexico City, Mexico City, Mexico
- Puerto Rico (2):
  - Akero Clinical Study Site, Manatí
  - Akero Clinical Study Site, San Juan
- South Korea (7):
  - Akero Clinical Study Site, Daegu, Daegu Gwang'yeogsi
  - Akero Clinical Study Site, Goyang-si, Gyeonggi-do
  - Akero Clinical Study Site, Incheon, Gyeonggi-do
  - Akero Clinical Study Site, Seongnam-si, Gyeonggi-do
  - Akero Clinical Study Site, Daegu, Gyeongsangbuk-do
  - Akero Clinical Study Site, Seoul, Seoul Teugbyeolsi [Seoul-T'ukpyolshi]
  - Akero Clinical Study Site, Seoul, Seoul Teugbyeolsi
- Switzerland (3):
  - Akero Clinical Study Site, Olten, Canton of Solothurn
  - Akero Clinical Study Site, Bern
  - Akero Clinical Study Site, Sankt Gallen
- Taiwan (4):
  - Akero Clinical Study Site, Changhua, Changhua
  - Akero Clinical Study Site, Taichung, Taichung
  - Akero Clinical Study Site, Tainan, Tainan
  - Akero Clinical Study Site, Taipei
- Turkey (Türkiye) (4):
  - Akero Clinical Study Site, Yenimahalle, Ankara
  - Akero Clinical Study Site, Bornova, İzmir
  - Akero Clinical Study Site, Bursa
  - Akero Clinical Study Site, Rize
- United Kingdom (3):
  - Akero Clinical Study Site, Liverpool, England
  - Akero Clinical Study Site, London, England
  - Akero Clinical Study Site, Newcastle upon Tyne, England

IPD SHARING:
Plan to Share IPD: No